CLINICAL TRIAL: NCT01478425
Title: Study on the Efficacy and Tolerability of a Topical Microemulsion in Patients With Intermittent or Persistent Allergic Rhinitis Due to Sensitization to Birch, Olive Tree or Grass Pollen
Brief Title: Efficacy and Tolerability of a Topical Microemulsion in Patients With Allergic Rhinitis Due to Sensitization to Pollen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reig Jofre Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RJ-NME-11-01
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Allergic Rhinitis
Keywords: Prevention; Pollen; Allergy; Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity; Rhinitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Lipidic Microemulsion
  Interventions: Device: Lipidic Microemulsion
- Control (Placebo Comparator): Saline nose-spray device
  Interventions: Device: Saline

INTERVENTIONS:
Device: Lipidic Microemulsion — Topical nasal, twice a day
  Other Names: Blox4
  Arms: Active
Device: Saline — Topical Nasal, twice a day
  Arms: Control

SUMMARY:
Study design: Randomized, controlled, double-blind, parallel, multicentre multinational clinical trial, to show superiority of an active therapy as compared to a control therapy on intermittent or persistent Allergic Rhinitis.

Primary objective:

1. To show that a topical microemulsion is superior to a sterilized saline solution to prevent deterioration in the health related quality of life, in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.

   Secondary objectives
2. To explore the effect of a topical microemulsion, as compared to a sterilized saline solution, for the prevention of nasal and ocular symptoms in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.
3. To explore the effect of a topical microemulsion, as compared to a sterilized saline solution, in the utilization of symptomatic medications, in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.
4. To assess the patient's satisfaction with a topical microemulsion treatment, as compared to a sterilized saline solution, in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.
5. To assess the safety of a topical microemulsion, as compared to a sterilized saline solution, administered to patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.

This is a clinical investigation study of a Class 1 medical device product. This is a prospective study of an active medical device versus a control medical device.

It was considered feasible to recruit 10 patients patients per center, and therefore the study should be conducted in 10 centers. To get treatment balance within each center, a total of 100 patients should be recruited.

DETAILED DESCRIPTION:
Main study investigator:

Dr. Pedro Ojeda Clínica de Asma y Alergia doctores Ojeda C/ Oquendo, 23 28006 Madrid, Spain T1.: +34 91 562 32 62 T2.: +34 91 562 67 27 F.: +34 91 562 53 96 e-mail: drojeda@telefonica.net

Objectives

Primary objective

1. To show that a topical microemulsion is superior to a sterilized saline solution to prevent deterioration in the health related quality of life, in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.

   Secondary objectives
2. To explore the effect of a topical microemulsion, as compared to a sterilized saline solution, for the prevention of nasal and ocular symptoms in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.
3. To explore the effect of a topical microemulsion, as compared to a sterilized saline solution, in the utilization of symptomatic medications, in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.
4. To assess the patient's satisfaction with a topical microemulsion treatment, as compared to a sterilized saline solution, in patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.
5. To assess the safety of a topical microemulsion, as compared to a sterilized saline solution, administered to patients with intermittent or persistent allergic rhinitis due to sensitization to birch, olive tree or grass pollen.

Study design:

Randomized, controlled, double-blind, parallel, multicentre multinational clinical trial, to show superiority of an active therapy as compared to a control therapy.

Study disease:

Intermittent or persistent Allergic Rhinitis.

Data from the drugs/interventions to be studied:

This is a clinical investigation study of a Class 1 medical device product. This is a prospective study of an active medical device versus a control medical device.

Study population and total number of subjects:

It was considered feasible to recruit 10 patients patients per center, and therefore the study should be conducted in 10 centers. To get treatment balance within each center, a total of 100 patients should be recruited.

In order to participate in the study, eligible candidates must fulfill all the following inclusion criteria and none of the exclusion criteria:

Inclusion criteria

1. Patients of either gender, aged 18 years or older.
2. With previous diagnostic of allergic rhinitis or rhinoconjunctivitis due to sensitization to birch, grass or olive tree pollens. Patients sensitized to other inhaled allergens might be included provided that these other sensitizations are not relevant to the patient's clinical symptoms or they are not exposed to these other allergens.
3. Having suffered from allergic rhinitis symptoms (severe enough to require symptomatic medication usually prescribed for this condition) in previous years, but otherwise free of symptoms at inclusion.
4. Residing during the months from March to July of 2011 in a geographical area in which the exposure to birch, grass or olive tree pollens is relevant (average pollination peaks of 100 grains/m3 of air during the previous specific pollen season).
5. Providing written informed consent to participate in the study.

Exclusion criteria

1. Known asthma of any origin (intrinsic or extrinsic, the latter due to any kind of allergenic trigger).
2. Allergic rhinitis or rhinoconjunctivitis whose symptoms are exclusively due to the sensitization to other inhaled allergens different from those referred in the inclusion criteria, sensitization to pollens that may interfere with the patient's allergic status during the study period (e.g., plane tree pollen).
3. Rhinitis or rhinoconjunctivitis of allergic characteristics presenting in the spring season but with negative allergy study (skin prick tests (SPT)).
4. Asymptomatic sensitization to birch, grass or olive tree pollens.
5. Sensitization to birch, grass or olive tree pollens, but having had mild symptoms during the spring of 2010, not requiring the use of symptomatic medication.
6. Sensitization to birch, grass or olive tree pollens but only presenting with asthma symptoms.
7. Concurrent participation in another clinical trial at the time of this study.
8. Co-morbid conditions that, in the investigator's judgment, preclude them from participating in this study.
9. Continuous treatment with antihistamines, corticosteroids, immunosuppressants or any other drug that may alter the occurrence and/or severity of allergic symptoms.
10. Individuals that, even if they meet the inclusion criteria, are concurrently under treatment with allergen-specific immunotherapy or have received this treatment within the last 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender, aged 18 years or older.
2. With previous diagnostic of allergic rhinitis or rhinoconjunctivitis due to sensitization to birch, grass or olive tree pollens. Patients sensitized to other inhaled allergens might be included provided that these other sensitizations are not relevant to the patient's clinical symptoms or they are not exposed to these other allergens.
3. Having suffered from allergic rhinitis symptoms (severe enough to require symptomatic medication usually prescribed for this condition) in previous years, but otherwise free of symptoms at inclusion.
4. Residing during the months from March to July of 2011 in a geographical area in which the exposure to birch, grass or olive tree pollens is relevant (average pollination peaks of 100 grains/m3 of air during the previous specific pollen season).
5. Providing written informed consent to participate in the study.

Exclusion Criteria:

1. Known asthma of any origin (intrinsic or extrinsic, the latter due to any kind of allergenic trigger).
2. Allergic rhinitis or rhinoconjunctivitis whose symptoms are exclusively due to the sensitization to other inhaled allergens different from those referred in the inclusion criteria, sensitization to pollens that may interfere with the patient's allergic status during the study period (e.g., plane tree pollen).
3. Rhinitis or rhinoconjunctivitis of allergic characteristics presenting in the spring season but with negative allergy study (skin prick tests (SPT)).
4. Asymptomatic sensitization to birch, grass or olive tree pollens.
5. Sensitization to birch, grass or olive tree pollens, but having had mild symptoms during the spring of 2010, not requiring the use of symptomatic medication.
6. Sensitization to birch, grass or olive tree pollens but only presenting with asthma symptoms.
7. Concurrent participation in another clinical trial at the time of this study.
8. Co-morbid conditions that, in the investigator's judgment, preclude them from participating in this study.
9. Continuous treatment with antihistamines, corticosteroids, immunosuppressants or any other drug that may alter the occurrence and/or severity of allergic symptoms.
10. Individuals that, even if they meet the inclusion criteria, are concurrently under treatment with allergen-specific immunotherapy or have received this treatment within the last 36 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
global score of the mini-RQLQ at visit 2 (adjusting for the baseline value)
  The primary analysis will be conducted on the global score of the mini-RQLQ at visit 2 (adjusting for the baseline value). It will be conducted on all randomized patients and will be considered as confirmatory. When visit 2 assessments are lacking, then no change from baseline will be assumed and baseline values will be carried forward to visit 2. As Normality and homcedasticity may be assumed, the analysis will consist of an ANCOVA model with a fixed treatment effect and baseline values as covariates.

SECONDARY OUTCOMES:
• Mini-RQLQ dimensions scores at visit 2
  Same analysis applied to the primary outcome but to individual dimensions of the RQLQ instead of global score
Mini-RQLQ global and dimensions scores at visit 3
  Same analysis applied to the primary outcome but to individual dimensions of the RQLQ instead of global score
Mean of the sums of nasal symptom scores at visits 2 and 3
  Same analysis applied to the primary outcome but to sums of nasal symptom scores at visits 2 and 3 instead of global score
Mean of the sums of ocular symptom scores at visits 2 and 3
  Same analysis applied to the primary outcome but to sums of ocular symptom scores at visits 2 and 3 instead of global score
Mean of the sums of symptomatic treatments at visits 2 and 3
  Same analysis applied to the primary outcome but to sums of symptomatic treatments at visits 2 and 3 instead of global score

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ojeda, PhD, MD, Study Director — Clínica Ojeda; Morgan Andersson, PhD, MD, Principal Investigator — Lund University Hospital; Julio Delgado, PhD, MD, Principal Investigator — Hospital Universitario Virgen Macarena; Ana Navarro, PhD, MD, Principal Investigator — Area Hospitalaria de Valme; Javier Subiza, PhD, MD, Principal Investigator — Clinica Subiza; José María Olaguibel, PhD, MD, Principal Investigator — Complejo Hospitalario de Navarra; Francisco Feo-Brito, PhD, MD, Principal Investigator — Hospital General de Ciudad Real; Juan Manuel Igea, PhD, MD, Principal Investigator — Clínica Alergoasma; Alicia Alonso, PhD, MD, Principal Investigator — Paracelso Clínica Médico Quirúrgica
Locations (9):
- Spain (8):
  - Hospital General de Ciudad Real, Ciudad Real, Ciudad Real
  - Clinica Ojeda, Madrid, Madrid
  - Clinica Subiza, Madrid, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Clinica Alergoasma, Salamanca, Salamanca
  - Hospital Universitario Virgen de la Macarena, Seville, Sevilla
  - Area Hospitalaria de Valme, Seville, Sevilla
  - Paracelso Clínica Médico Quirúrgica, Valladolid, Valladolid
- Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Ojeda P, Pique N, Alonso A, Delgado J, Feo F, Igea JM, Navarro A, Olaguibel JM, Subiza J, Nieto C, Andersson M. A topical microemulsion for the prevention of allergic rhinitis symptoms: results of a randomized, controlled, double-blind, parallel group, multicentre, multinational clinical trial (Nares study). Allergy Asthma Clin Immunol. 2013 Aug 27;9(1):32. doi: 10.1186/1710-1492-9-32. PMID 23981504